CLINICAL TRIAL: NCT00090454
Title: Genetic Markers of CHD Risk in Men and Women
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Richard P Donahue, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 1266; R01HL075389 (NIH)
Record Dates: First submitted 2004-08-26; First posted 2004-08-30 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2008-07

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Inflammation

SUMMARY:
To investigate the association of selected genetic markers of inflammation and endothelial activation with the occurrence of non-fatal acute myocardial infarction (MI).

DETAILED DESCRIPTION:
BACKGROUND:

Coronary artery disease is a major cause of death and disability in westernized societies, and is growing in importance in countries with emerging economies. Inflammation and endothelial dysfunction are now recognized as important contributors to coronary artery disease. However, the genetic basis and specific genes involved in the expression of the hyperinflammatory phenotype are not yet well-understood. Identification and further characterization of variation in candidate loci that are associated with coronary artery disease would contribute to the understanding of the genetic basis underlying acute myocardial infarction, and may provide novel pathways for prevention and treatment.

DESIGN NARRATIVE:

This case-control study will determine whether the variability in several genes that influence inflammation and endothelial dysfunction is related to the odds of myocardial infarction (MI) among 700 men and 229 postmenopausal women from the Western New York Health Study. The study performs the following: 1) To test the hypothesis that cases of acute MI will have a higher frequency of specific haplotypes at the C-reactive protein locus composed of alleles associated with higher levels of CRP production (-732G/A), 1059G/C, and +1444C/T) than matched controls. MI cases will have a greater frequency of haplotypes composed of alleles associated with higher levels of interleukin (IL) production, specifically IL-6 production (-597G/A, -572G/C, and -174G/C) than controls, and a lower frequency of specific haplotypes in the IL1A/IL1 BILL1RN gene region; 2) cases will have a higher frequency of alleles and haplotypes for specific functional polymorphisms of the E-selectin gene (128R and G98T) than controls; 3) to utilize DNA pooling strategy for rapid screening of large numbers of single nucleotide polymorphisms (SNPs) in 29 candidate genes in relevant biological pathways and test selected loci for association with risk of acute MI; 4) for those loci with evidence of association, to identify haplotype tagging single nucleotide polymorphisms (htSNPs) that capture the variation at each locus and test for association between these SNPs and haplotypes and risk of MI. Secondary aims will a) explore the above associations among men with premature MI (55 years of age or less) and b) explore gene- gene and gene- environment interactions. MI case subjects were identified from hospital record review in Erie and Niagara counties (95% of all eligible cases, ICD9 410-410.9) an average of 4 months post MI. They were interviewed and examined in 1996-2001. Control subjects were randomly selected from the same counties (59.5% response rate) and had a contemporaneous clinical exam. Controls will be individually matched to cases by age, sex, and ethnicity.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Donahue — State University of New York at Buffalo